CLINICAL TRIAL: NCT00296803
Title: PROCLAIM: Pilot Study Examining Effects of Clopidogrel Compared to Placebo on Markers of Inflammation in Subjects With Metabolic Syndrome
Brief Title: PROCLAIM: Study Examining Effects of Clopidogrel Compared to Placebo on Inflammation in Subjects With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_9842
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Metabolic Syndrome x
Keywords: metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Clopidogrel

INTERVENTIONS:
Drug: clopidogrel

SUMMARY:
The purpose of this study is to examine the effects of clopidogrel compared to placebo on markers of inflammation in subjects with metabolic syndrome who are receiving background therapy including low dose aspirin.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years old
2. Women must be post-menopausal for one year, surgically sterilized, or using a medically accepted method of contraception and must agree to use an effective method of contraception throughout the study.
3. Subject must meet 3 of the 5 National Cholesterol Education Program/Adult Treatment Panel III (NCEP/ATP III) criteria for the classification of metabolic syndrome: triglycerides >/= 150 mg/dL; blood pressure (BP): systolic blood pressure (SBP) >/= 130 mmHg/diastolic blood pressure (DBP) > 85 mmHg; fasting glucose >/= 110 mg/dL; waist circumference: men - > 101.6 cm (40 in)/women - > 88.9 cm (35 in); high-density lipoprotein (HDL) cholesterol: men - < 40 mg/dL/women - < 50 mg/dL.
4. Subject has high-sensitivity C-reactive protein (hs-CRP) levels of >/= 2.0 but <10.0 mg/L at the Screening Visit (Week -2).
5. Current medication regimen must be stable for six (6) weeks, i.e. no initiation of new prescription medication nor change in dosage of any previously initiated medication within three months of entering this study.
6. Subject is normally active and judged to be in good health, based on medical history, routine safety laboratory tests (Screening Visit, Week -2), and a brief physical examination (Week -2).

Exclusion Criteria:

1. Intolerance or contraindication to the use of clopidogrel or aspirin.
2. Thrombocytopenia as defined by platelet count < 100,000/mm3.
3. Current use or use within the past 3 months of oral anticoagulants, or dipyridamole or thienopyridine (ticlopidine or open-label clopidogrel) or oral glucocorticoids.
4. Daily aspirin in excess of 81 mg, or chronic use of non-steroidal anti-inflammatory agents.
5. Use of oral hormone replacement therapy or oral contraceptives including transdermal patch.
6. History of pathologic bleeding (i.e., peptic ulcer or intracranial hemorrhage).
7. History of chronic inflammatory disease or any recent medical event(s) resulting in tissue injury, infection, or inflammation.
8. Myocardial infarction, coronary artery bypass graft, or angioplasty within the 6 months prior to Screening.
9. Uncontrolled hypertension (systolic blood pressure >/= 180 mmHg or diastolic blood pressure >/= 100 mmHg) at Screening.
10. History or presence of cancer in the past 2 years, except for successfully resected basal cell carcinoma of the skin.
11. Recent history (within the past 12 months) for alcohol or substance abuse.
12. Currently taking another investigational study medication or has taken investigational study medication within 30 days prior to Screening Visit.
13. Any condition the Investigator believes would interfere with evaluation of the subject, or which could put the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216
Dates: Start 2005-11; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To assess the effects of clopidogrel + aspirin vs placebo + aspirin on hs-CRP, CD40-ligand, soluble P-selectin, and other selected biomarkers in subjects with metabolic syndrome and elevated hs-CRP levels at study baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lilienthal, M.S., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States